CLINICAL TRIAL: NCT01020526
Title: A 6-month, Open-label, Safety Trial Of Pregabalin In Adolescent Patients With Fibromyalgia
Brief Title: Pregabalin In Adolescent Patients With Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A0081231; 2010-020300-29 (EudraCT Number)
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Results first posted 2016-07-01 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2016-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pregabalin (Experimental)
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — Oral capsule 75-450 mg/day

SUMMARY:
The main purpose of this study is to evaluate the long-term safety of pregabalin in adolescent patients who participated in the previous fibromyalgia study (A0081180) and who wish to recieve open-label pregabalin

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met the inclusion criteria for the preceding fibromyalgia Study A0081180, and have received pregabalin/placebo under double-blind conditions.

Exclusion Criteria:

* Patients may not participate in the study if they experienced a serious adverse event during the previous fibromyalgia study A0081180 which was determined to be related to the study medication by the investigator or sponsor.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2010-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (21):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Apex Research Institute, Santa Ana, California
  - Florida Medical Center & Research, Miami, Florida
  - Harmony Clinical Research, Incorporated, North Miami Beach, Florida
  - Rheumatology Associates of Central Florida, PA, Orlando, Florida
  - Medical Research & Health Education Foundation, Inc., Columbus, Georgia
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - University Pediatric Rheumatology of Kentucky, LLC, Louisville, Kentucky
  - University of Massachusetts Memorial Medical Center Department of Pediatrics, Worcester, Massachusetts
  - Akron Children's Hospital, Akron, Ohio
  - Akron Children's Hospital-Mahoning Valley, Boardman, Ohio
  - Akron Children's Hospital, Boardman, Ohio
  - University of Cincinnati Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Medical University of South Carolina, Pediatric Rheumatology, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Carolina Research Center, Myrtle Beach, South Carolina
  - Fatigue Consultation Clinic, Salt Lake City, Utah
- Bioregeneracni a rehabilitacni centrum, Říčany, Czechia
- India (4):
  - Krishna Institute of Medical Sciences Ltd, Secunderabad, Andhra Pradesh
  - Mallikatta Neuro Center, Mangalore, Karnataka
  - Sushrut Hospital, Research Centre & Post Graduate Institute of Orthopaedics, Nagpur, Maharashtra
  - King George's Medical University, Lucknow, Uttar Pradesh

REFERENCES:
- [Derived] Arnold LM, Schikler KN, Bateman L, Khan T, Pauer L, Bhadra-Brown P, Clair A, Chew ML, Scavone J; Pregabalin Adolescent Fibromyalgia Study Group. Safety and efficacy of pregabalin in adolescents with fibromyalgia: a randomized, double-blind, placebo-controlled trial and a 6-month open-label extension study. Pediatr Rheumatol Online J. 2016 Jul 30;14(1):46. doi: 10.1186/s12969-016-0106-4. PMID 27475753
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081231&StudyName=Pregabalin%20In%20Adolescent%20Patients%20With%20Fibromyalgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 63 participants were screened and enrolled at 19 study centers in this open-label extension study to the parent double-blind randomized fibromyalgia study A0081180.
Groups:
- Pregabalin: Participants initiated dosing at 75 mg/day and their dose was optimized over a 3 week period, based on tolerability and response, to a dose of 75 mg/day, 150 mg/day, 300 mg/day or 450 mg/day. These doses were administered during the subsequent flexible dosing phase for a period of 21 weeks. Pregabalin was administered orally as capsules.
Period: Overall Study
Arm/Group | Pregabalin
Started | 63
Completed | 49
Not Completed | 14
Not completed — Withdrawal by Subject | 5
Not completed — Other reasons | 3
Not completed — Insufficient clinical response | 3
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.8 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Numeric Rating Scale by Week
Description: The weekly pain numeric rating scale (Weekly Pain NRS) consists of an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicate worse pain. Participants chose the number that best described the pain during the last week. Negative change indicates improvement.
Time Frame: Baseline, Weeks 3, 8, 16, 24 and Last Visit.
Population: This population will include all participants who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Number
Arm/Group | Pregabalin
Number analyzed (Participants) | 63
Number
  Baseline (N=63) | 6.7 (1.68)
  Week 3 (N=61) | -2.1 (2.51)
  Week 8 (N=55) | -1.8 (2.95)
  Week 16 (N=51) | -2.1 (2.6)
  Week 24 (N=55) | -2.1 (2.56)
  Last Visit (N=63) | -2.1 (2.47)

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from the time the participants had taken at least one dose of study drug through the last subject visit.
Description: For summary purposes, adverse event investigator terms were converted to preferred terms using a standard system of classification (COSTART or MedDRA). Adverse events tabulations included summaries by body system or system organ class, by overall decreasing frequency and by maximum intensity.
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 3/63
Other Adverse Events (participants affected / at risk) | 32/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=63)
Appendicitis (Infections and infestations) | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1
Migraine (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pregabalin (N=63)
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Ear infection (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Dizziness (Nervous system disorders) | 14
Headache (Nervous system disorders) | 6
Dysmenorrhoea (Reproductive system and breast disorders) | 3/53 — The number of females is 53 out of 63 participants and dysmenorrhoea occurs in females only thus exceeds 5%.
Fatigue (General disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study participating sites. Investigator may not disclose previously undisclosed confidential other than study results.